CLINICAL TRIAL: NCT04431648
Title: Novel MRI-Guided Ultrasound Stimulated Microbubble Radiation Treatment for Patients With Head and Neck Cancer
Acronym: USmBRT-H
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Gregory Czarnota, Senior Scientist, MD, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 076-2019
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer; Focused Ultrasound; Microbubble
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — perflutren

STUDY DESIGN:
Intervention Model Description: Prospective, Single-Centre, Single-Arm, Non-Randomized, Phase-I MRI-Guided Ultrasound Stimulated Microbubbles Radiation Treatment for Patients with Head and Neck Cancers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRg-FUS MB Treatment (Experimental): Patients with head and neck cancer will receive MRI-guided ultrasound-stimulated microbubble-treatment combined with radiotherapy on a LINAC.
  Interventions: Drug: DEFINITY; Device: Sonalleve Focused Ultrasound Device

INTERVENTIONS:
Drug: DEFINITY — MRI-guided ultrasound-stimulated microbubble-treatment
Device: Sonalleve Focused Ultrasound Device — Sonalleve Focused Ultrasound Device

SUMMARY:
The objective of this study is to demonstrate the feasibility of novel MRI-guided ultrasound stimulated microbubble treatment to enhance radiation effects in humans receiving external beam radiotherapy delivered using a LINAC (linear accelerator) radiation therapy device.

DETAILED DESCRIPTION:
This study is to demonstrate the feasibility of novel MRI-guided ultrasound stimulated microbubble treatment to enhance radiation effects in humans receiving external beam radiotherapy delivered using a LINAC (linear accelerator) radiation therapy device. The investigators have previously demonstrated that ultrasound and microbubble mediated endothelial cell perturbation can significantly enhance the effectiveness of radiation. It enhances tumour response to radiation significantly by synergistically destroying tumour blood vessels. The technique is targeted spatially and achieves tumour specificity by confining the low-power ultrasonic fields that stimulate microbubbles to the tumour location only. By perturbing the tumour vasculature and activating specific genetic pathways, the technique sensitizes the targeted tissues to the subsequent therapeutic application of radiation, resulting in significantly enhanced cell killing. The primary aim of this research is to evaluate the safety profile of MRI-guided ultrasound stimulated microbubble treatment and radiation in patients with head and neck cancer. The secondary aim is to evaluate tumor (primary and/or nodal) response to MRg-FU + MB and radiation, as measured radiologically within the treated therapeutic regions.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* All biopsy-confirmed squamous cell carcinoma (SCC) of the H&N including the following subregions: Larynx, Oropharynx, Hypopharynx, Oral Cavity, Salivary Glands, and Paranasal Sinuses
* Stage I-IV H&N cancers (i.e. cT1-T4, cN0-N3, cM0), per AJCC guidelines (8th Edition).
* Assessed by the treating surgeon, and radiation oncologist, and following a multidisciplinary discussion, determined to have unresectable and/or inoperable disease in the head and neck region.
* Patients referred for palliative radiotherapy or standard radiotherapy, including the following dose regimens: 70 Gy/35 fractions, 50 Gy/20 fractions, or 35-40 Gy/5 fractions (SBRT, hypofractionation).
* Patients treated with concurrent pre-operative chemoradiation, including: Cisplatin (40 mg/m2 q.w.k or Carboplatin 70 mg/m2 / day IV on days 1-4, 22-25 and at days 43-46 of radiation) or referred for palliative radiotherapy.
* Able to understand and give informed consent.
* Weight <140kg.
* Radiologic evidence of neck lymphadenopathy with at least one target lesion measuring > 1cm in largest dimension (Recurrent or initial presentation)
* Target lesion visible by non-contrast MRI.
* Target lesion accessible for MRg-FU procedure.
* Able to communicate sensation during MRg-FU treatment.
* Creatinine within normal institutional limits or creatinine clearance >60 mL/min/1.73 m2 for patients with creatinine levels above institutional upper limit of normal

Exclusion Criteria:

* Pregnant or lactating women may not participate due to the embryotoxic effects of protocol treatment. Women/ men of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.
* Unable to have contrast-enhanced MRI scan - standard of care criteria
* Head and neck surgery (excluding biopsy) ≤ 6 weeks prior to study enrolment
* Chemotherapy or other systemic anti-cancer agents ≤ 1 week prior to enrolment unless cisplatin-based chemotherapy
* Previous radiotherapy ≤ 6 weeks prior to enrollment
* Target lesion involves the skin surface causing ulceration, bleeding or discharge
* Target lesion in contact with hollow viscera
* Target lesion located in the skull, spine, or mandible
* The fibrotic scar along the proposed FU beam path
* Orthopedic implant along proposed FU beam path or at a site of the target lesion.
* Severe cardiovascular, neurological, renal or hematological chronic disease
* ECOG (Eastern Cooperative Oncology Group) Performance Status ≥ 3. Unable to tolerate required stationary position during treatment
* Cardiac disease or unstable hemodynamics including myocardial infarction within six months, unstable angina, congestive heart failure, ejection fraction < 50%, cardiac shunts, cardiac arrythmia and cardiac pacemaker.
* Contraindication to perflutren including subjects with a family or personal history of QT prolongation or taking concomitant medications known to cause QTc prolongation like cisapride, erythromycin, tricyclic antidepressants, Class IA and III antiarrhythmic agents and some antipsychotics like haloperidol, droperidol, quetiapine, thioridazine, ziprasidone. QT prolongation observed on screening ECG (QTc > 450ms for men or >470ms for women)
* Severe hypertension (diastolic BP > 100 mmHg)
* History of bleeding disorder, coagulopathy
* Severely impaired renal function with estimated glomerular filtration rate < 30ml/min/1.73m2 and/or on dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of toxicity and adverse events using MRg-FUS MB treatment in patients with head and neck cancer | 90 days
  Incidence of toxicity and adverse events

SECONDARY OUTCOMES:
Radiological response | 90 days
  The secondary endpoint is radiological response in head and neck cancer following MRg-FU + MB + radiation, after a 3 month follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory J Czarnota, PhD, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Gregory J Czarnota, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No